CLINICAL TRIAL: NCT03347747
Title: Asymmetrical Facial Volume Loss From Disproportionate Light Exposure: A Clinical Validation Study
Brief Title: Facial Asymmetrical Clinical Evaluation Study
Acronym: FACE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: McDaniel Institute of Anti-Aging Research (Industry)
Collaborators: Allergan (Industry); Merz Aesthetics Inc. (Industry); ThermiGen, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: FCLVOL-2017
Record Dates: First submitted 2017-11-05; First posted 2017-11-20 (Actual); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Loss of Facial Adipose Tissue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Photoaged Male Subjects: 45-80 year old males with visible photoaging and the desired exposure profile/driving history and who also has spent (or are spending) at least 30 minutes in a car per day (as the driver), 5 days per week for at least 15 years of their adult life to ensure they have the type of asymmetrical exposure required for hypothesis validation. This is an multi-center trial, and study sites will range from northern to southern latitudes in North America, Australia and potentially other international sites. Study Photography + Personal & Medical History Collection via a study questionnaire will be obtained.
  Interventions: Other: Study Photography + Personal & Medical History Collection
- Photoaged Female Subjects: 45-80 year old females with visible photoaging and the desired exposure profile/driving history and who also has spent (or are spending) at least 30 minutes in a car per day (as the driver), 5 days per week for at least 15 years of their adult life to ensure they have the type of asymmetrical exposure required for hypothesis validation. This is an multi-center trial, and study sites will range from northern to southern latitudes in North America, Australia and potentially other international sites. Study Photography + Personal & Medical History Collection via a study questionnaire will be obtained.
  Interventions: Other: Study Photography + Personal & Medical History Collection

INTERVENTIONS:
Other: Study Photography + Personal & Medical History Collection — 3D facial images taken and complete a detailed study questionnaire

SUMMARY:
The primary objective of this study is to create digital 3D images of subjects using a Canfield VECTRA H1 digital imaging system and compile a medical, skin/sun exposure and sunscreen use, and skin care product history for a large number of subjects. This data will allow for image and statistical analysis to determine if facial volume loss is greater on one side, and what factors may be causing this.

The data collected will also serve as a database for future lines of inquiry relating to data collected in this study. Your data (including 3D images) will be kept in this database and may be accessed in the future by any Sponsor or Investigator. Your data will be de-identified and your name will not be associated with the questionnaire responses

DETAILED DESCRIPTION:
It has been long noted that facial volume loss is one of the primary visible components of aging. Asymmetrical volume loss has been noted as well, but there is no proven theory explaining why this occurs.

This study will attempt to determine whether there is an association between greater facial volume loss on the drivers' window side of the face.

This data will allow for image and statistical analysis to determine if a facial volume loss differential exists, and what factors may be isolated to determine causality The study population will be between 350-500 males or females aged 45-80 having visible photodamage and spent (or are spending) at least 30 minutes in a car per day (as the driver), 5 days per week for at least 15 years of their adult life to ensure they have the type of asymmetrical exposure required for hypothesis validation.

This will be a multi-center trial, and study sites will range from northern to southern latitudes in North America, Australia and potentially other international sites.

This study is to be conducted under the general supervision of PI(s) and will follow the general guidelines recommended in current Good Clinical Practices (cGCP).

Individual sites will have a PI to supervise study related procedures and data collection and will be in contact with Dr. McDaniel and staff throughout the study.

The study period for each subject will be approximately 1-2 visits. Consented and qualified subjects will be imaged using the Canfield VECTRA H1 digital imaging system as described above and then given the study questionnaire and completion instructions. Once the subject has had both the images and questionnaire reviewed by study personnel for completeness, their participation in this study is ended; unless the supplemental contact visit is determined to be required for data clarification or additional, IRB approved, follow up questions.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 45 to 80 years of age with no known medical conditions that, in the investigator's opinion, may interfere with study participation.

  2. Subjects must have spent, at minimum, an average of at least 30 minutes per day/ 5 days per week (as the driver) in an automobile for greater than or equal to 15 years of their adult life.

  3. Subjects must sign a written informed consent. 4. Subjects must agree to be photographed with the 3D camera system and sign a photo release.

  5. Subjects must agree to fill out the study questionnaire completely and to the best of their knowledge.

  6. Subjects must agree that the de-identified data and 3D images may be used for data mining to answer future study questions or assist in new investigations and discoveries.

Exclusion Criteria:

* Any dermatologic disorder, which in the investigator's opinion, may interfere with the accurate evaluation of the subject's facial skin. Examples of such disorders include severe acne vulgaris, acne conglobata, acne fulminans, facial seborrheic dermatitis, and lupus erythematosus.

  2. Concurrent therapy with any medication either topical or oral that might, in the investigator's opinion, interfere with the study.

  3. Subjects who have had performed procedures which, in the study doctor's opinion, may interfere with the study data (for example: face lift, facial liposuction or facial volume fillers in the last 2 years) 4. Subjects whose primary automobile (used in the average drive estimate) has dark tinted window glass or UV filter applied to the driver's side window glass.

  5. Subjects who have spent a large portion of their lives at two very different latitude/locations (eg. Alternate 6 months of the year at a summer home in Maine and a winter home in Florida).

  6. Subjects who are unwilling or unable to comply with the requirements of the protocol.

  7. Subject has any disorder that may prevent compliance, such as history of chronic alcohol or drug abuse, significant mental or nervous disorder or other illness that would, in the evaluator's opinion, interfere with the study.

  8. Subjects with visible (or excessive vellus) facial hair (facial hair interferes with the 3D imaging capture and analysis).

  9. Subject's weight has ever been more than 30 lbs above or below current weight (does not include weight gain associated with pregnancy)

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: the study will consist of up to 500 volunteer 45-80 year old males or females with visible photoaging and the desired exposure profile/driving history. If a subject meets study criteria and is enrolled, they will have 3D facial images taken and complete a detailed study questionnaire
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2017-06-09 (Actual); Primary Completion 2018-06-30 (Estimated); Study Completion 2018-07-31 (Estimated)

PRIMARY OUTCOMES:
Study Photos and Questionnaire Data Processing | June 2018
  The questionnaire data will be entered into a central spreadsheet for future analysis. The images will be uploaded directly to Canfield Scientific for image review and analyzed using software based on a "best fit" algorithm designed using 1000 facial images to determine any volume differences between the right and left sides of the face. Statistical significance will be generated for the data and applied to the general population of 300,000,000 with a 95% confidence interval (based on a study population of 400 subjects). Detailed statistics may be performed utilized using an online statistics calculator as required. The full complement of images and data from each site, will be returned to the McDaniel Institute of Anti-Aging Research.

CONTACTS AND LOCATIONS:
Overall Officials: Daivd H. McDaniel, MD, Study Director — MIAAR
Locations (1):
- McDaniel Institute of Anti-Aging Research, Virginia Beach, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided